CLINICAL TRIAL: NCT01432782
Title: Prospective Randomised Double-blind Sham Study on the Use of Botox for the Treatment of Diffuse Esophageal Spasm
Brief Title: Botulinum Toxin Injection to Treat Diffuse Esophageal Spasm
Acronym: Botox
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Prof Dr Jan Tack, Professor of Medicine, Universitaire Ziekenhuizen KU Leuven
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BotoxDES
Record Dates: First submitted 2011-09-09; First posted 2011-09-13 (Estimated); Last update posted 2011-09-13 (Estimated); Status verified 2011-09

CONDITIONS: Esophageal Spasm, Diffuse
Keywords: Weight loss; Dysphagia; Esophageal hypermotility; Chest Pain
MeSH Terms: conditions — Esophageal Spasm, Diffuse; Weight Loss; Deglutition Disorders; Chest Pain | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo arm: per-endoscopic injection of saline
  Interventions: Drug: Placebo
- Botulinum toxin (Active Comparator): Botulinum toxin (Botox) 100 u in 4 ml, injected per-endoscopically
  Interventions: Drug: Botulinum Toxin Type A

INTERVENTIONS:
Drug: Placebo — Saline 4 ml
  Arms: Placebo
Drug: Botulinum Toxin Type A — per-endoscopic injection of 100 U of botulinum toxin dissolved in 4 ml of saline
  Other Names: Botox
  Arms: Botulinum toxin

SUMMARY:
This study evaluates the effect of botulinum toxin 100 U or saline, injected endoscopically in the distal esophagus, on symptoms and manometry pattern in patients with diffuse esophageal spasm.

DETAILED DESCRIPTION:
Patients are selected on the basis of a clinical diagnosis of diffuse esophageal spasm, based on endoscopy and manometry.

This is a sham-controlled cross-over study of injection of botulinum toxin or saline, in randomized order, in the distal esophagus.

All patients have undergone esophageal manometry which shows diffuse esophageal spasm, and a 24h pH monitoring/manometry to quantify acid reflux. All drugs prescribed to affect esophageal motility (nitrates, calcium antagonists) are stopped during the study. After randomisation, the patient will undergo standard esophageal manometry to assess baseline esophageal motility. On the same day the patient will be asked to fill out a set of symptom questionnaires including a dysphagia questionnaire. At endoscopy, the active treatment group receives 8 x 12.5 units, each in 0.5 ml, of botulinum toxin A which will be injected in the four quadrants of the esophagus at 2 and 5 cm above the lower esophageal sphincter. In the Sham group 8 * 0.5 ml of physiologic serum will be injected. The randomisation will be performed at the endoscopy unit by a nurse otherwise not involved in the protocol.

After 1 month a stationary manometry and a new esophageal pH/manometry monitoring will be performed, followed by a second endoscopy with injection of saline or botulinum toxin in a cross-over mode. At the time of the second endoscopy each patient will fill out a dysphagia questionnaire. One month later, the dysphagia questionnaire is repeated.

Subsequently, follow-up will occur at the outpatient clinic after 6 and 12 months, with follow-up dysphagia questionnaires but no additional manometries or endoscopies, unless the clinical status deteriorates.

ELIGIBILITY:
Inclusion Criteria:

* Spastic motor disorder in the upper GI tract

Exclusion Criteria:

-

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-02; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Dysphagia severity score | One month after treatment
  the primary outcome variable is the symptom severity score in patients with diffuse esophageal spasm.

SECONDARY OUTCOMES:
Manometry pattern | One month after treatment
  Pattern of contractions on stationary esophageal manometry

CONTACTS AND LOCATIONS:
Overall Officials: Jan Tack, M.D., Ph.D., Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- University Hospitals Leuven, Leuven, Flanders, Belgium